CLINICAL TRIAL: NCT01627158
Title: Pharmacokinetic Study Comparing Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler Forte; a Randomised, Double-blind, Double-dummy, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Study Comparing Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler Forte
Acronym: ADECO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3103011
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Charcoal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide/formoterol Easyhaler (Experimental): Budesonide/formoterol Easyhaler
  Interventions: Drug: Budesonide/formoterol Easyhaler
- Symbicort Turbuhaler (Active Comparator): Symbicort Turbuhaler
  Interventions: Drug: Symbicort Turbuhaler
- Charcoal and Budesonide/formoterol Easyhaler (Experimental)
  Interventions: Drug: Charcoal and Budesonide/formoterol Easyhaler
- Charcoal and Symbicort Turbuhaler (Active Comparator)
  Interventions: Drug: Charcoal and Symbicort Turbuhaler

INTERVENTIONS:
Drug: Budesonide/formoterol Easyhaler — Budesonide/formoterol Easyhaler
  Arms: Budesonide/formoterol Easyhaler
Drug: Symbicort Turbuhaler — Symbicort Turbuhaler
  Arms: Symbicort Turbuhaler
Drug: Charcoal and Budesonide/formoterol Easyhaler — Charcoal and Budesonide/formoterol Easyhaler
  Arms: Charcoal and Budesonide/formoterol Easyhaler
Drug: Charcoal and Symbicort Turbuhaler — Charcoal and Symbicort Turbuhaler
  Arms: Charcoal and Symbicort Turbuhaler

SUMMARY:
The purpose of this study is to compare the test product Budesonide/formoterol Easyhaler with the marketed product Symbicort Turbuhaler in terms of the drug absorbed into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Males and females, 18-60 (inclusive) years of age.

Exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
2. Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of study results or constitute a health risk for the subject if he/she takes part in the study.
3. Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
4. Known hypersensitivity to the active substance(s) or the excipient of the drug.
5. Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax of plasma budesonide concentration | within 12 h
Pharmacokinetic parameter AUCt of plasma budesonide concentration | 12 h
Pharmacokinetic parameter Cmax of plasma formoterol concentration | 24 h
Pharmacokinetic parameter AUCt of plasma formoterol concentration | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Irja Korpela, MSc, Study Director — Orion Corporation, Orion Pharma; Rainard Fuhr, Dr. med., Principal Investigator — Parexel Berlin
Locations (1):
- PAREXEL International GmbH, Berlin, Germany